CLINICAL TRIAL: NCT06303024
Title: Targeting Subclinical Motor and Cognitive Impairment in Patients With Early Onset Multiple Sclerosis at High Risk of disEase Acitivity Through a Preventive personaLised and InnovAtive rehaBiLitation stratEgy. (RELIABLE)
Brief Title: Targeting Subclinical Motor and Cognitive Impairment in Patients With Early Onset Multiple Sclerosis
Acronym: RELIABLE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Collaborators: Careggi Hospital (Other); Sheba Medical Center (Other Government); Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RELIABLE Clinical Study
Record Dates: First submitted 2024-03-04; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-02

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting

STUDY DESIGN:
Intervention Model Description: This is a multicentric no-profit pilot study, composed by two phases. I phase: observational prospective study II phase: interventional study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- personalized combined physical and cognitive intervention (Experimental): The exercise intervention will be aerobic and performed on a stationary bicycle and will comply with the basic principle of progressive overload, combined with a computer based cognitive rehabilitation program carried out twice a week for 12 weeks, using the Rehacom software.
  Interventions: Other: personalized combined physical and cognitive intervention

INTERVENTIONS:
Other: personalized combined physical and cognitive intervention — The exercise intervention will be aerobic and performed on a stationary bicycle and will comply with the basic principle of progressive overload. An incremental exercise test until exhaustion on a bicycle ergometer will be applied to determine directly measured VO2-max in order to customize and personalize the training on each patient. The progressive aerobic exercise (PAE) will last 12 weeks with two sessions per week. Continuous training will be alternated with interval training during the program. The intervention included two weekly training sessions. One session will involve continuous exercise initially commencing at 10 min and progressing towards 30 min/session. Ultimately, a computer based cognitive rehabilitation program will be carried out twice a week for 12 weeks, using the Rehacom software. Participants will begin at level 1 on each RehaCom module and advance through the program as dictated by their performance. Each session will be programmed to last 60 minutes.

SUMMARY:
Our project proposal is based on an individualized rehabilitation approach in patients with early stage relapsing remission (RR) MS. This approach will be based on risk stratification obtained using several clinical and demographic parameters that are not commonly used in clinical practice. This risk score will be obtained from an extensive neuropsychological, psychosocial and physical assessment to which patients will undergo at baseline and at one-year follow-up.The risk score will allow a better stratification of patients' risk of disease worsening/progression and the application of a preventive and personalized strategy.

DETAILED DESCRIPTION:
This is a multicentric no-profit pilot study, composed by two phases. The objective of the first phase is to create a multi-factorial assessment and prognostic profiling into different risk categories, integrating different techniques in a common evaluation approach. MS patients, referred to the MS Centers of Careggi University Hospital and the Sheba Medical Centre in Tel-Aviv, will be recruit and assess at baseline and 12-months follow-up using a comprehensive approach. The patients will undergo an advanced motor performance evaluation, neuropsychological assessment, and a brain MRI scan to evaluate the presence of new/enlarging T2 lesions, new gadolinium-positive lesions, and volumetric analyses (e.g., total brain volume, grey matter volume, white matter volume, T2 lesions volume, normalized thalamic and hippocampal volume). Data collected from the comprehensive baseline and 12 months assessment will be used to generate a risk score for disease worsening in the short-term, classifying the patients into low/mild, moderate, or high risk. All the variables significantly associated with disease activity will be combined in the risk score.The objectives of II Phase are to apply the previously obtained risk score on a novel cohort using the same inclusion/exclusion criteria; to evaluate the impact of a combined rehabilitation approach in reducing the proportion of patients with disease activity.The risk score obtained from follow-up data of the test cohort applied to the newly recruited patients. Only patients with moderate to high risk of worsening in this new cohort will be included in the rehabilitation program. The included patients will receive an innovative and personalized rehabilitation approach, including counselling on lifestyle habits, an aerobic moderate to high-intensity physical training and a computerized cognitive rehabilitation program.The efficacy of the rehabilitation approach will be then evaluated by comparing patients included in this cohort with patients in the same risk groups included in the phase 1 cohort. Across Phases of the study, Uppsala University partner, will conduct a surveillance and will consider Social and ethical aspects of the integrated rehabilitation approach. Personalized preventive interventions and tailored risk information may raise pressing ethical issues that need careful reflection.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of RRMS based on the 2017 McDonald criteria;
* age ≥ 18 years;
* EDSS ≤ 2.0;
* disease duration ≤ 5 years;
* verification of MS subtype,
* duration of disease and EDSS will be accomplished by obtaining a signed consent form for the release of medical information from the treating neurologist.

Exclusion Criteria:

* history of relevant psychiatric comorbidities.
* Severely depressed subjects assessed through the Beck Depression Inventory (scores ≥ 29);
* relapses or corticosteroid treatment in the 30 days before inclusion;
* history of substance abuse;
* presence of non-MS related physical or cognitive impairment that could make the patient unable to complete the study assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2023-06-14 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Symbol Digit Modalities Test (SDMT) | baseline and 1 year followup cohort 1; baseline, 3 months and 1 year followup cohort 2
  The SDMT is a simple matching task that requires the participant to refer to a reference key, in order to correctly match a geometric symbol with the corresponding number. Participant will be under a 90 second time constraint to quickly and correctly match each pair.
California Verbal Learning Test second edition (CVLT-II) | baseline and 1year followup cohort 1; baseline, 3 months and 1year followup cohort 2
  The CVLT test begins with the examiner reading a list of 16 words, participants are then instructed to report as many of the words as they can remember. After recall is recorded, the entire list is read again, altogether, there are five learning trials.
Brief Visuo-Spatial Memory Test- Revised (BVMT-R) | baseline and 1 year followup cohort 1; baseline, 3 months and 1year followup cohort 2
  Participants are presented with six abstract designs for 10 seconds, the display is then removed from view and participant are instructed to draw the designs from memory via pencil on paper. Each design is scored from 0 to 2 points representing accuracy and location. There are three learning trials.
Word list generation (WLG) | baseline and 1year followup cohort 1; baseline, 3 months and 1year followup cohort 2
  the subject has to say as many words from the fruit and vegetable categories as they can think of in one and a half minutes
Stroop test | baseline and 1year followup cohort 1; baseline, 3 months and 1year followup cohort 2
  the reading time of the stimuli in the interference condition is assessed: there are colours written but the colour of the ink is different from the written word, the subject has to say the colour of the ink in which the word is written
Test Intelligenza Breve (TIB) | baseline cohort 1 and baseline cohort 2
  evaluation of the IQ estimation, the subject reads words with regular and irregular accents and takes the number of errors of words with irregular accents
9 hole peg test (9HPT) | baseline and 1year followup cohort 1; baseline, 3 months and 1year followup cohort 2
  to measure finger dexterity, the subject must take the pegs one at a time with the dominant hand and then with the other hand and insert them as quickly as possible into the holes and remove them
The Hospital Anxiety and Depression Scale (HADS) | baseline and 1year followup cohort 1; baseline, 3 months and 1 year followup cohort 2
  to measure anxiety and depression
Beck Depression Inventory second edition | baseline and 1year followup cohort 1; baseline, end 3 months and 1year followup cohort 2
  to measure depression
The Modified Fatigue Impact Scale (MFIS) | baseline and 1year followup cohort 1; baseline, 3 months and 1year followup cohort 2
  to measure fatigue
The Multiple Sclerosis Walking Scale (MSWS-12) | baseline and 1year followup cohort 1; baseline, 3 months and 1year followup cohort 2
  evaluate the participants subjective impact of walking.
Multiple Sclerosis Impact Scale (MSIS-29-V2) | baseline and 1yearfollowup cohort 1; baseline, 3 months and 1year followup cohort 2
  to evaluate the participants impact of Multiple Sclerosis.
Multiple Sclerosis Quality of Life-54 (MSQOL-54) | baseline and 1year followup cohort 1; baseline, 3 months and 1year followup cohort 2
  to evaluate quality of life
six minutes walking test (6MWT) | baseline and 1year followup cohort 1; baseline, 3 months and 1year followup cohort 2
  to measure the distance a subject can travel by walking as fast as possible on a flat surface in six minutes.
Romberg test | baseline and 1year followup cohort 1; baseline, 3 months and 1year followup cohort 2
  to assess balance
handgrip test | baseline and 1year followup cohort 1; baseline, 3 months and 1year followup cohort 2
  a strength evaluation test
cognitive-motor interference | baseline and 1year followup cohort 1; baseline, 3 months and 1year followup cohort 2
  impact of a simple cognitive test - verbal fluency on a randomly extracted letter - on motor performances
Timed 25-foot walk | baseline and 1year followup cohort 1; baseline, 3 months and 1year followup cohort 2
  is a quantitative mobility and leg function performance test based on a timed 25-walk.
brain MRI scan | baseline and 1 year followup cohort 1 and 2
  to evaluate the presence of new/enlarging T2 lesions, new gadolinium-positive lesions, and volumetric analyses
International Physical Activity Questionnaire (IPAQ) | baseline and 1 year followup cohort 1 and 2
  to assess the types of intensity of physical activity and sitting time that people do as part of their daily lives are considered to estimate total physical activity in MET-min/week and time spent sitting.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Fondazione Don Carlo Gnocchi ONLUS, Florence, Italy

IPD SHARING:
Plan to Share IPD: No